CLINICAL TRIAL: NCT00552786
Title: Antioxidation Medication for Noise-induced Hearing Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Institute of Occupational Safety and Health, Taiwan (Unknown); Municipal Hospital of Tainan, Taiwan (Unknown)
Responsible Party: Dr. Yue-Liang Guo, National Taiwan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 200704018M
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Results first posted 2010-07-27 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2009-11

CONDITIONS: Hearing Loss
Keywords: noise; hearing loss; temporary threshold shift
MeSH Terms: conditions — Hearing Loss | interventions — Acetylcysteine; Glucose; Sugars

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetin (Experimental)
  Interventions: Drug: N-acetylcysteine (NAC)
- Glucose (Placebo Comparator)
  Interventions: Drug: glucose

INTERVENTIONS:
Drug: N-acetylcysteine (NAC) — 600mg twice daily for 2 weeks
  Other Names: acetin (600mg)
  Arms: Acetin
Drug: glucose — 1 gm glucose capsule
  Other Names: Sugar
  Arms: Glucose

SUMMARY:
This study will examine whether oral intake of 1200mg N-Acetylcysteine/day will prevent temporary threshold shift in hearing among workers exposed to noise

DETAILED DESCRIPTION:
Both genetic and environmental factors contribute to noise-induced hearing loss (NIHL). The cellular antioxidant system appears to protect cochlear hair cells from oxidative stress due to noise. Previous animal studies showed protective effects of anti-oxidant medicines against NIHL.The objective of this study is to test the hypothesis that preventive medication of antioxidation is related to susceptibility to NIHL.

The 53 noise-exposed workers from steel industries in Taiwan will be recruited, and divided into N-Acetylcysteine (NAC)(Acetine, 1200mg/day) group and placebo one. The duration of medication is 2 weeks initially. After washout for 2 weeks, the kinds of medications in these 2 groups will be crossover and used for 2 weeks. Firstly, questionnaires interview about noise exposure, smoking, alcohol drinking, drug habit history and calculation of Body Mass Index (BMI) will be done. The following methods would be performed individually after medication. With detailed local examination with otoscope, these subjects receive hearing tests by pure-tone audiometry (PTA) and distortion product otoacoustic emissions (DPOAE) before and after their daily works. The possible confounding factors including background noise, solvent, heavy metals, carbon monoxide and temperature in the workplaces will be assessed. The amount of noise exposure is evaluated by personal dosimeter. Early morning, Blood samples will be collected. Deletion polymorphisms in the Glutathione S-transferase (GST)T1 and GSTM1 genes will be determined. Statistical analysis will be performed to evaluate the relation between intake of anti-oxidant medicine and noise-induced temporal threshold shift (TTS).

The expected results of this study are to determine whether anti-oxidant supplements protect workers from noise-induced TTS.

We anticipate that these human studies might help elucidate the relative importance of anti-oxidant enzymes as risk factors for NIHL.

ELIGIBILITY:
Inclusion Criteria:

* workers in steel industry
* known exposure to noise at work

Exclusion Criteria:

* ever diagnosed as having diabetes mellitus
* fasting glucose of 120 or greater

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yue-Liang L Guo, MD, MPH, PHD, Principal Investigator — National Taiwan University Hospital; Tung-Sheng Shih, PHD, Study Director — Institute of Occupational Safety and Health, Taiwan
Locations (1):
- Environmental and Occupational Medicine, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Coleman JK, Kopke RD, Liu J, Ge X, Harper EA, Jones GE, Cater TL, Jackson RL. Pharmacological rescue of noise induced hearing loss using N-acetylcysteine and acetyl-L-carnitine. Hear Res. 2007 Apr;226(1-2):104-13. doi: 10.1016/j.heares.2006.08.008. Epub 2006 Oct 4. PMID 17023129
- [Background] Kopke R, Bielefeld E, Liu J, Zheng J, Jackson R, Henderson D, Coleman JK. Prevention of impulse noise-induced hearing loss with antioxidants. Acta Otolaryngol. 2005 Mar;125(3):235-43. doi: 10.1080/00016480410023038. PMID 15966690
- [Background] Duan M, Qiu J, Laurell G, Olofsson A, Counter SA, Borg E. Dose and time-dependent protection of the antioxidant N-L-acetylcysteine against impulse noise trauma. Hear Res. 2004 Jun;192(1-2):1-9. doi: 10.1016/j.heares.2004.02.005. PMID 15157958
- [Background] Kopke RD, Jackson RL, Coleman JK, Liu J, Bielefeld EC, Balough BJ. NAC for noise: from the bench top to the clinic. Hear Res. 2007 Apr;226(1-2):114-25. doi: 10.1016/j.heares.2006.10.008. Epub 2006 Dec 20. PMID 17184943
- [Derived] Lin CY, Wu JL, Shih TS, Tsai PJ, Sun YM, Ma MC, Guo YL. N-Acetyl-cysteine against noise-induced temporary threshold shift in male workers. Hear Res. 2010 Oct 1;269(1-2):42-7. doi: 10.1016/j.heares.2010.07.005. Epub 2010 Jul 16. PMID 20638463

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between November 2007 and January 2008.
Pre-assignment Details: A total of 60 workers voluntarily participated in this study. However, 6 workers had preexisting hearing loss of >50 dBA at high frequency and 1 worker accidentally turned off the noise monitoring device. These 7 participants were excluded from the analysis. The 53 workers who satisfactorily completed the study.
Groups:
- N-acetylcysteine (NAC) First, Then Placebo: Formulation NAC (1200 mg/day, 14 days) (Actein, Synmosa Corp., Taiwan) in the first intervention period and Placebo (a tablet of identical taste and odor to the NAC agent) in the second intervention period (after washout period).
- Placebo First, Then N-acetylcysteine (NAC): Placebo in the first intervention period and Formulation NAC in the second intervention period (after washout period).
Period: First Intervention
Arm/Group | N-acetylcysteine (NAC) First, Then Placebo | Placebo First, Then N-acetylcysteine (NAC)
Started | 25 | 28
Medication and Hearing Evaluation | 25 | 28
Completed | 25 | 28
Not Completed | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | N-acetylcysteine (NAC) First, Then Placebo | Placebo First, Then N-acetylcysteine (NAC)
Started | 25 | 28
Completed | 25 | 28
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | N-acetylcysteine (NAC) First, Then Placebo | Placebo First, Then N-acetylcysteine (NAC)
Started | 25 | 28
Completed | 25 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetylcysteine (NAC) First, Then Placebo | Placebo First, Then N-acetylcysteine (NAC) | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 25 | 28 | 53.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.0 (11.6) | 42.1 (9.6) | 41.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0.0
  Male | 25 | 28 | 53.0
Region of Enrollment [Number; unit: participants]
  Taiwan | 25 | 28 | 53.0

OUTCOME MEASURES:

1. Primary Outcome: Temporary Threshold Shift Measurement by Pure Tone Audiometry (A Total of Four Hearing Assessments Were Completed for Each Formulation Period on the 1st Day Pre- and Post-shift, and the 14th Day Pre- and Post-shift)
Description: The hearing threshold level (HL) at high frequency (HF) by pure-tone audiometry (PTA) was defined as the average of HLs at 3k,4k,6kHz for each ear examined. A total of four hearing assessments by PTA were completed for each formulation period on the 1st day pre- and post-shift, and the 14th day pre- and post-shift. The amount of temporary threshold change was calculated by subtracting the pre-shift hearing threshold from the post-shift hearing threshold at each frequency.
Time Frame: A total of four hearing assessments were completed for each formulation period on the 1st day pre- and post-shift, and the 14th day pre- and post-shift
Population: Intent to treat analysis including only participants who had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: decibels
Groups:
- N-acetylcysteine (NAC): Formulation NAC (1200 mg/day, 14 days) (Actein, Synmosa Corp., Taiwan) administered in either first intervention period or second intervention period.
- Placebo: Placebo administered once daily in either first intervention period or second intervention period.
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 53 | 53
decibels | 3.4 (2.3) | 2.7 (2.1)
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA — Two-sided; Assessing the bioequivalence on temporary threshold shift at3k,4k,6k Hz between NAC and Placebo was carried out using ANOVA for 2×2 crossover design

2. Secondary Outcome: Temporary Threshold Changes Measurement by Distortion Product Otoacoustic Emissions (DPOAE) (A Total of Four Hearing Assessments Were Completed for Each Formulation Period on the 1st Day Pre- and Post-shift, and the 14th Day Pre- and Post-shift)
Description: Distortion product otoacoustic emissions (DPOAE) is an objective measure to assess the cochlear changes. DPOAE response threshold at high frequency (HF) was defined as the average of response levels (dB SPL) at 3k,4k,6kHz for each ear examined. A total of four hearing assessments by DPOAE were completed for each formulation period on the 1st day pre- and post-shift, and the 14th day pre- and post-shift. The amount of DPOAE temporary threshold change was calculated by subtracting the pre-shift DPOAE response threshold from the post-shift DPOAE response threshold at each frequency.
Time Frame: as for outcome 1
Population: Intent to treat analysis including only participants who had all 4 post-baseline assessments (measurements at beginning of 1st and 2nd intervention periods and end of 1st and 2nd intervention periods).
Measure: Mean (Standard Deviation); unit: decibels (dB SPL)
Arm/Group | N-acetylcysteine (NAC) | Placebo
Number analyzed (Participants) | 53 | 53
decibels (dB SPL) | -0.85 (1.1) | -0.89 (0.9)
Statistical Analysis 1: Comparison: N-acetylcysteine (NAC) vs Placebo; Test type: Superiority or Other; p < 0.05, ANOVA; Assessing the bioequivalence on temporary threshold shift at 3k,4k,6k Hz between NAC and Placebo was carried out using ANOVA for 2×2 crossover design

ADVERSE EVENTS:
Arm/Group | N-acetylcysteine (NAC) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

LIMITATIONS AND CAVEATS:
No text entered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No